CLINICAL TRIAL: NCT04183699
Title: Identifying the Optimal Biopsy Scheme at MRI Target Biopsy
Brief Title: Optimizing the Number of Systematic COres During a MRI Target Biopsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Prof. Alberto Briganti, Full Professor, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SCOT
Record Dates: First submitted 2019-11-07; First posted 2019-12-03 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Suspicion of Prostate Cancer With a Positive Multiparametric Magnetic Resonance of the Prostate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI targeted + systematic random biopsy (Experimental)
  Interventions: Diagnostic Test: Prostate biopsy

INTERVENTIONS:
Diagnostic Test: Prostate biopsy — MRI-targeted + systematic random prostate biopsy

SUMMARY:
This is a multicentre, paired-cohort, prospective, controlled study. The patient with a suspicion of PCa and a concomitant positive mpMRI (defined as presence of one lesion PI-RADS ≥ 3) will receive a MRI-TBx (4 target cores). During the same session, subsequently to MRI-TBx, patient will receive a systematic sampling with 6-core S-Bx followed by 14-core S-Bx, for a total of 20-core systematic cores, in addition to 4 MRI-TBx cores. Procedure will be performed by the same operator. Each single core will be stored in a dedicated cassette and sequentially numbered. We hypothesize that the proportion of csPCa (defined as prostate cancer with Gleason score ≥ 3+4) detected by 6-cores S-Bx will be no less than that detected by 20-cores S-Bx, both performed in addition to MRI-TBx. Assessing the optimal number of systematic cores to take in addition to MRI-TBx cores in men undergoing a MRI-TBx would provide a useful clinical information for every day clinical practice. Moreover, the possibility to decrease the number of systematic cores taken during a MRI-TBx, hence reducing the overall number of cores taken during a biopsy, would reduce the length of the diagnostic procedure, potentially reduce the probability of infections/sepsis and reduce the overdiagnosis of clinically insignificant PCa.

ELIGIBILITY:
Inclusion Criteria:

* Male patients, aged between 18 and 80 years old with suspicion of prostate cancer
* Presence of a positive mpMRI of the prostate (visible lesion PI-RADS ≥ 3)
* Serum PSA ≤ 20ng/ml
* Suspected stage ≤ T2 on rectal examination (organ confined prostate)
* Fit to undergo a prostate biopsy
* Able to understand and willing to sign a written informed consent document

Exclusion Criteria:

* Prior positive prostate biopsy
* Prior treatment of the prostate
* Prostate volume <30 ml at mpMRI of the prostate
* More than one lesion at mpMRI of the prostate
* Contraindication to prostate biopsy

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Estimated)
Dates: Start 2019-06-06 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Detection rate of clinically significant prostate cancer with 6-core vs. 20-core systematic biopsy during a MRI target biopsy | through study completion, an average of 1 year
  Proportion of patients diagnosed with csPCa with 6-core vs. 20-core systematic biopsy during a MRI target biopsy

SECONDARY OUTCOMES:
Incremental value of any additional systematic and targeted core on the detection rate of clinically significant prostate cancer during MRI target biopsy | through study completion, an average of 1 year
  The proportion of men diagnosed with csPCa according to the addition of any single systematic core

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele, Milan, Italy